CLINICAL TRIAL: NCT01238432
Title: The Genetics of Severe Asthma in Children
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: UConn Health (Other)
Responsible Party: Sponsor
Other Study IDs: 08-103
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2022-10

CONDITIONS: Asthma
Keywords: Pediatric; Polymorphism, Genetic; Adrenergic beta-Agonists
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inpatient population: Children with asthma who are admitted to the hospital with an exacerbation.
- Outpatient population: Children with asthma who have not been admitted to the hospital with an exacerbation.
- Healthy controls: Children without asthma or any other chronic condition.

SUMMARY:
Near fatal asthma exacerbations are one of the most common causes of critical illness in children, accounting for approximately ten thousand intensive care unit (ICU) admissions per year in the United States. Even children with intermittent or mild baseline asthma can develop these severe exacerbations; however, there are few studies evaluating the risk factors associated with the development of near fatal asthma exacerbations in children. Inhaled β2-adrenergic receptor (ADRβ2) agonist therapy is the foundation of therapy for acute asthma and genetic variations of this receptor have been shown to affect response to ADRβ2 agonist therapy in this population. The investigators hypothesis is that a child's ADRβ2 genotype is associated with the development of a near fatal asthma exacerbation.

DETAILED DESCRIPTION:
Our primary outcome measure is the development of a near fatal asthma exacerbation. Secondary outcome measures will include the duration of continuously nebulized ADRβ2 agonist therapy and the duration of IV ADRβ2 agonist therapy. Children will be stratified by ADRβ2 genotype at amino acid position 16 and outcomes compared.

We propose to investigate two separate populations in this study: (1) children admitted to the hospital with an acute asthma exacerbation, and (2) children with asthma who have never had an acute near fatal asthma exacerbation. In addition, in order to replicate findings in an independent cohort, we will examine the genotypes of a third cohort of age-matched children without asthma.

For the population of children admitted to the hospital with an acute asthma exacerbation, the following inclusion criteria will be met: (1) admission to the hospital with a primary admission diagnosis of asthma exacerbation and (2) age between 4 years and 18 years. Near fatal asthma exacerbations will be defined as (1) treatment with intubation and mechanical ventilation, (2) presence of respiratory acidosis (arterial pCO2 > 45), or (3) Modified Pulmonary Index Score > 12 after 2 hours of at least 20 mg/hour of continuously nebulized albuterol therapy. Children will be excluded if they have a (1) pre-existing chronic disease (other than asthma) including: (a) bronchopulmonary dysplasia, (b) bronchomalacia, (c) tracheomalacia, (d) laryngomalacia, (e) vocal cord dysfunction, (f) chronic restrictive lung disease, (g) recurrent aspiration pneumonia, or (h) congenital heart disease.

For the population of children with asthma who have never had an acute near fatal asthma exacerbation, the following inclusion criteria will be met: (1) diagnosis of asthma and (2) age between 4 years and 18 years. Children will be excluded if (1) that child ever required admission to the hospital for a near fatal asthma exacerbation and (2) if they have a pre-existing chronic disease (other than asthma) as listed above. We propose to enroll 158 children, recruited from Pulmonary Clinic at the study institution, matched by age, by gender, and by NHLBI asthma classification to the population of children with near fatal asthma exacerbations.

In order to replicate these findings in an independent cohort, we will also examine these genetic markers in a reference group of 80 healthy children without asthma, matched by age, gender and race/ethnicity to the group of children with near fatal asthma exacerbations. The following inclusion criteria will be met for this group: (1) age between 4 and 18 years. Children will be excluded if they have any pre-existing chronic disease. This population of children will be recruited from the Primary Care Clinic at CCMC and if necessary for racial/ethnic matching, from a private practice in suburban Hartford.

For the population of children hospitalized with an asthma exacerbation, patients will be approached, consented and enrolled upon admission to the hospital. In this observational study, patients will be treated according to the current asthma treatment protocol in effect at Connecticut Children's Medical Center. This protocol has been previously published 13 and titrates therapy based on a clinical asthma score (MPIS) 51 that has been shown to be highly reproducible between groups of physicians, nurses and respiratory therapists. This around-the-clock adjustment of therapy by nurses and respiratory therapists produces less variation in care due to non-medical reasons. This protocol includes thresholds for admission/discharge to the hospital and for admission/discharge to the ICU based on MPIS. For the populations of children with no history of a near fatal asthma exacerbation and no asthma diagnosis, patients will be approached, consented and enrolled upon confirmation of eligibility in the Pulmonary Clinic and the Primary Care Clinic.

Genotyping of the ADRβ2 gene will be performed at the University of Connecticut Health Center (UCHC) Clinical and Translational Research Core Lab. Genotyping will be performed either from saliva or from whole blood collected during routine blood sampling for clinical care. Children will be stratified based on their genotype and outcomes compared. Providers will be blinded to genotype at the time of treatment.

ELIGIBILITY:
Inclusion Criteria, inpatient asthmatics:

* Admission to study institution with a primary admission diagnosis of asthma exacerbation
* Age between 4 and 18 years

Exclusion Criteria, inpatient asthmatics:

- Pre-existing chronic disease (other than asthma), including: i. bronchopulmonary dysplasia ii. bronchomalacia iii. tracheomalacia iv. laryngomalacia v. vocal cord dysfunction vi. chronic restrictive lung disease vii. recurrent aspiration pneumonia viii. impaired mucous clearance ix. congenital heart disease x. pulmonary hypertension

Inclusion Criteria, outpatient asthmatics:

* Diagnosis of asthma
* Age between 4 and 18 years

Exclusion Criteria, outpatient asthmatics:

* Previous admission to the hospital for a near fatal asthma exacerbation
* Pre-existing chronic disease (other than asthma) including i. bronchopulmonary dysplasia ii. bronchomalacia iii. tracheomalacia iv. laryngomalacia v. vocal cord dysfunction vi. chronic restrictive lung disease vii. recurrent aspiration pneumonia viii. impaired mucous clearance ix. congenital heart disease x. pulmonary hypertension

Inclusion Criteria, healthy controls:

- Age between 4 and 18 years

Exclusion Criteria, healthy controls:

- Pre-existing chronic disease including: i. asthma ii. bronchopulmonary dysplasia iii. bronchomalacia iv. tracheomalacia v. laryngomalacia vi. vocal cord dysfunction vii. chronic restrictive lung disease viii. recurrent aspiration pneumonia ix. impaired mucous clearance x. congenital heart disease xi. pulmonary hypertension

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with asthma
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2009-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The primary end point is the development of a near fatal asthma exacerbation. | 3 years

SECONDARY OUTCOMES:
The secondary end point is hospital length of stay. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Carroll, MD, MS, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No